CLINICAL TRIAL: NCT04917328
Title: Evaluation of the Predictive Value of Compression Venous Ultrasound by the Emergency Physician for Excluding the Diagnosis of Proximal Deep Vein Thrombosis (DVT) in Patients With Non-high Clinical Pretest Probability
Brief Title: Compression Ultrasonography in Non-high Probability of Deep Vein Thrombosis
Acronym: EPREVUP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8114
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with clinical suspicion of deep vein thrombosis (Experimental)
  Interventions: Other: compression ultrasound

INTERVENTIONS:
Other: compression ultrasound — performing a compression ultrasound

SUMMARY:
Compression ultrasound is commonly used in emergency department. Accuracy to rule out deep vein thrombosis is excellent but lower then Ddimer assessment which is actually gold standard. With progress in formation of emergency physicians (EP), quality of material used, the investigators hypothesize that compression ultrasound can rule out deep vein thrombosis in case of non high probability, as standard care and DDimer assay.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* Patient presenting to the emergency department with clinical suspicion of DVT (i.e. pain and/or lower extremity edema).
* Patient with a non-high probability according to the modified Wells score, i.e. a score of 0 or 1
* Subject with a social health insurance plan
* Subject able to understand the objectives and risks of the research and to give a signed and dated informed consent

Exclusion Criteria:

* Patient with suspected pulmonary embolism
* Patient with a high probability of DVT
* Impossible to perform a whole leg doppler ultrasound within 5 days
* Pregnant or breast-feeding woman, on patient's declaration
* Subject under court protection
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value of compression ultrasound for diagnosis of deep vein thrombosis | The measurement is assessed during ED stay or in 5 days if DD is positive with no DVT in compression ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Strasbourg, Strasbourg, France